CLINICAL TRIAL: NCT04462848
Title: Phase I Study of the Safety and Pharmacokinetics of Human Convalescent Plasma in High Risk Children Exposed or Infected With SARS-CoV-2
Brief Title: Covid-19 Convalescent Plasma as Prevention and Treatment for Children With Underlying Medical Conditions
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Jaime G. Deville, MD, FAAP, Clinical Professor of Pediatrics, University of California, Los Angeles
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB#20-001263
Record Dates: First submitted 2020-06-30; First posted 2020-07-08 (Actual); Last update posted 2020-07-08 (Actual); Status verified 2020-07

CONDITIONS: Corona Virus Infection
MeSH Terms: conditions — Coronavirus Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- anti-SARS-CoV-2 human convalescent plasma (Experimental): single transfusion of human convalescent plasma
  Interventions: Biological: anti-SARS-CoV-2 human convalescent plasma

INTERVENTIONS:
Biological: anti-SARS-CoV-2 human convalescent plasma — Single transfusion. The total volume (mL) to be transfused will be based on participant weight (kg) and will be calculated as 5 mL/kg. The maximum volume to be transfused will be 500 mL.

SUMMARY:
This study will provide access to investigational anti-SARS-CoV-2 human convalescent plasma for pediatric patients with underlying medical conditions (cardiovascular disease, lung disease, immunosuppression) who are either infected with SARS-CoV-2 or who have had a high-risk exposure. Study participants will be transfused once with compatible convalescent plasma obtained from an individual who has recovered from documented infection with SARS-CoV-2. Safety information and pharmacokinetic data will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 1 month and < 18 years at the time of consent.
* Determined to be at high-risk for severe SARS-CoV-2 disease based on the American Academy of Pediatrics definition of immunocompromised children and reported high-risk pediatric subpopulations. These include the following groups: immunocompromised, hemodynamically significant cardiac disease (e.g. congenital heart disease), lung disease with chronic respiratory failure, infant, i.e. child ≤1 year old.
* Confirmed SARS-CoV-2 infection OR high-risk exposure as defined:

  * Confirmed infection: Child who tested positive for COVID-19 and is no more than 96 hours after onset of symptoms (and within 120 hours at the time of receipt of study plasma).
  * High-risk exposure: Susceptible child who was not previously infected or otherwise immune to SARS-CoV-2 and exposed within 96 hours prior to enrollment (and within 120 hours at the time of receipt of study plasma). Both criteria below should be met:

    1. A household member or daycare center (same room) exposure to a person with confirmed SARS-CoV-2 OR with clinically compatible disease in areas with widespread ongoing transmission
    2. Negative for SARS-CoV-2 (nasopharyngeal or oropharyngeal swab)
* For females of reproductive potential (defined as having experienced menarche), not pregnant based on testing performed at screening.
* Parent or legal guardian able and willing to provide signed parent permission.

Exclusion Criteria:

* History of severe reactions (e.g. anaphylaxis) to transfusion of blood products. Individuals with minor reactions such as fever, itching, chills, etc. that resolve spontaneously or respond to pre-medications, and that do not represent more significant allergic reactions, will not be excluded.
* For females, breastfeeding, or planning to become pregnant/breastfeed during the study period.
* Participant is unlikely to adhere to the study procedures, keep appointments, or is planning to relocate outside the greater Los Angeles area during the study.
* Any condition that would, in the opinion of the principal investigator, place the participant at an unacceptable risk of injury or render the participant unable to meet the requirements of the protocol.

Ages: 1 Month to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2020-08 (Estimated); Primary Completion 2024-09 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Cumulative incidence of Grade 3 and Grade 4 adverse events | up to Day 28 post-administration of study plasma
  A Grade 3 adverse event is any untoward or unfavorable medical occurrence in which symptoms are severe and cause inability to perform usual social and functional activities with medical intervention or therapy indicated.
  A Grade 4 adverse event is any untoward or unfavorable medical occurrence in which potentially life-threatening symptoms cause inability to perform basic self-care functions with medical intervention or therapy indicated to prevent permanent impairment, persistent disability, or death.
Cumulative incidence of serious adverse events | up to Day 28 post-administration of study plasma
  A serious adverse event is any untoward or unfavorable medical occurrence that:
  * results in death,
  * is life-threatening,
  * requires inpatient hospitalization or prolongation of existing hospitalization,
  * results in persistent or significant disability/incapacity
  * is a congenital anomaly/birth defect, or
  * is an important medical event that may or may not be immediately life-threatening or result in death or hospitalization but may jeopardize the participant or may require intervention to prevent one of the other outcomes listed in the definition above.

SECONDARY OUTCOMES:
Proportion of participants with disease worsening event. | up to Day 28 post-administration of study plasma
  Descriptive analysis of disease worsening event as represented by hospitalization, prolongation of hospitalization, need for supplemental oxygen, respiratory distress, requirement for mechanical ventilation, and death.
Serum concentration at baseline, Day 7, Day 14, and Day 28 for anti-SARS-CoV-2 antibodies | Days 0, 7, 14, and 28
  Anti-SARS-CoV-2 antibody titer changes over time
Percentage of participants with a natural antibody response to SARS-CoV-2 infection | once between Day 60 and Day 120
  This will be assessed by the presence or absence of anti-SARS-CoV-2 antibody titers to be collected once between 60 and 120 days post study plasma administration

CONTACTS AND LOCATIONS:
Overall Officials: Jaime G Deville, M.D., Principal Investigator — UCLA Clinical Professor of Pediatrics
Locations (1):
- University of California, Los Angeles (UCLA), Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No